CLINICAL TRIAL: NCT00630955
Title: NMDA Antagonist Efficacy in Reducing Human Alcohol Consumption: Impact of Family History
Brief Title: Family History Study of Alcohol Consumption Using Memantine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0602001068; P50AA012870 (NIH)
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Drinking
Keywords: Alcohol Drinking; Memantine
MeSH Terms: conditions — Alcohol Drinking | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 20 mg memantine
  Interventions: Drug: memantine
- 2 (Experimental): 40 mg memantine
  Interventions: Drug: Memantine
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: memantine — Memantine 20 mg once per day for 7 days
  Other Names: Namenda
  Arms: 1
Drug: Memantine — Memantine 40 mg once per day for 7 days
  Other Names: Namenda
  Arms: 2
Drug: Placebo — Placebo once per day for 7 days
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effects of the study medication, memantine (placebo, 20 mg or 40 mg/day) on alcohol drinking behavior in a laboratory setting in which participants are given an initial drink of alcohol followed by the choice to drink up to 12 more drinks over a three-hour period. We hypothesize that memantine will reduce craving and number of drinks consumed prior to and after exposure to the initial drink of alcohol and during the three hour drinking period. We will also evaluate the influence of family history of alcoholism on the efficacy of memantine in reducing alcohol drinking behavior.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-50
* Able to read English at 6th grade level or higher and to complete study evaluations
* Regular alcohol drinker

Exclusion Criteria:

* Individuals who are seeking alcohol treatment
* Medical conditions that would contraindicate the use of memantine
* Regular use of other substances

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2006-06; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- CMHC, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://info.med.yale.edu/ctna/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2006-May 2011 using posted advertisements in the local newspaper and brochures and other materials distributed in the community (bars, coffee shops, grocery stores).Electronic media and social networking were also used, including Craigslist and Facebook.
Groups:
- 0 mg Memantine: Participants who received placebo PO qd
- 20 mg Memantine: Participants randomized to 20 mg memantine PO qd
- 40 mg Memantine: Participants randomized to 40mg memantine PO qd
Period: Overall Study
Arm/Group | 0 mg Memantine | 20 mg Memantine | 40 mg Memantine
Started | 34 | 37 | 40
Completed | 31 | 31 | 28
Not Completed | 3 | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0 mg Memantine | 20 mg Memantine | 40 mg Memantine | Total
Number analyzed (Participants) | 34 | 37 | 40 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 37 | 40 | 111
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (7.2) | 32.4 (9.3) | 31.3 (8.8) | 31.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 13 | 36
  Male | 23 | 25 | 27 | 75
Region of Enrollment [Number; unit: participants]
  United States | 34 | 37 | 40 | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Consumed on Day 7
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: standard drinks
Groups:
- 0 mg Memantine: Participants who received placebo
- 20 mg Memantine: Participants randomized to 20 mg memantine
- 40 mg Memantine: Participants randomized to 40mg memantine
Arm/Group | 0 mg Memantine | 20 mg Memantine | 40 mg Memantine
Number analyzed (Participants) | 31 | 31 | 28
standard drinks | 5.84 (3.67) | 5.61 (4.6) | 6.21 (4.61)

2. Primary Outcome: Baseline-adjusted Craving (YCS)
Description: Craving for alcohol based on Yale Craving Scale, scores ranging from 0-112 mm on a visual analog scale, with higher measurements indicating higher craving. The baseline-adjusted craving is change score from baseline at Day 7.
Time Frame: Day 7
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | 0 mg Memantine | 20 mg Memantine | 40 mg Memantine
Number analyzed (Participants) | 31 | 31 | 28
millimeters | 20.2 (2.16) | 14.1 (2.23) | 21.4 (2.23)

3. Secondary Outcome: Stimulation Responses to Alcohol
Description: Brief Biphasic Alcohol Effects Scale-Stimulation subscale, measuring stimulation effects of alcohol on Day 7, 6 items, 11-point rating scale from 0=Not at All to 10=Extremely, total scores ranging from 0 - 30, with higher measurements indicating higher stimulation.
Time Frame: Day 7
Population: Analysis includes all those who had complete data, which is less than those listed in the Participant Flow module
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0 mg Memantine | 20 mg Memantine | 40 mg Memantine
Number analyzed (Participants) | 28 | 28 | 27
units on a scale | 4.643 (4.923) | 4.321 (5.313) | 6.444 (6.536)

4. Secondary Outcome: Sedation Responses to Alcohol
Description: Brief Biphasic Alcohol Effects Scale-Sedation subscale, measuring sedation effects of alcohol on Day 7, 6 items, 11-point rating scale from 0=Not at All to 10=Extremely, total scores ranging from 0 - 30, with higher measurements indicating higher sedation.
Time Frame: Day 7
Population: Analysis includes all those who had complete data, which is less than those listed in the Participant Flow module
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0 mg Memantine | 20 mg Memantine | 40 mg Memantine
Number analyzed (Participants) | 28 | 28 | 27
units on a scale | 3.286 (5.381) | 3.964 (6.327) | 3.37 (5.085)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at baseline and during the 7 days of medication, as well as at the one week follow up
Groups:
- 0 mg: Participants who received placebo
- 20 mg: Participants randomized to 20 mg memantine
- 40 mg: Participants randomized to 40mg memantine
Arm/Group | 0 mg | 20 mg | 40 mg
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/37 | 0/40
Other Adverse Events (participants affected / at risk) | 22/34 | 24/37 | 31/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0 mg (N=34) | 20 mg (N=37) | 40 mg (N=40)
Abdominal Pain (Gastrointestinal disorders) | 6 | 2 | 3
nausea (Gastrointestinal disorders) | 9 | 5 | 10
vomit (Gastrointestinal disorders) | 5 | 2 | 0
Headache (General disorders) | 9 | 12 | 16
Dizzy (Nervous system disorders) | 5 | 3 | 12
fatigue (General disorders) | 6 | 5 | 9
nervous (Psychiatric disorders) | 3 | 4 | 0
insomnia (Nervous system disorders) | 2 | 4 | 7
confusion (Nervous system disorders) | 3 | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No